CLINICAL TRIAL: NCT03214094
Title: Special Drug Use Surveillance of Takecab Tablets for "Prevention of Recurrence of Gastric/Duodenal Ulcer in Patients Receiving Low-dose Aspirin: Long-term Use"
Brief Title: Special Drug Use Surveillance of Vonoprazan for "Prevention of Recurrence of Gastric/Duodenal Ulcer in Patients Receiving Low-dose Aspirin: Long-term Use"
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Vonoprazan-5004; JapicCTI-163435 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2017-07-09; First posted 2017-07-11 (Actual); Results first posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-02

CONDITIONS: Gastric or Duodenal Ulcers
MeSH Terms: conditions — Duodenal Ulcer | interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vonoprazan 10 mg: The usual adult dosage for oral use is 10 mg of Vonoprazan administered once daily. Participants will receive interventions as part of routine medical care.
  Interventions: Drug: Vonoprazan

INTERVENTIONS:
Drug: Vonoprazan — Vonoprazan tablets
  Other Names: Takecab tablets; TAK-438

SUMMARY:
The purpose of this survey is to investigate the safety and effectiveness of long-term administration of vonoprazan tablets for up to 12 months in the routine clinical setting in patients receiving low-dose aspirin.

DETAILED DESCRIPTION:
The drug being tested in this survey is called vonoprazan. Vonoprazan is being tested to treat people who have gastric or duodenal ulcers.

This survey will look at the safety and effectiveness of long-term administration of vonoprazan tablets for up to 12 months in the routine clinical setting in patients receiving low-dose aspirin.

The survey will enroll approximately 1,000 participants.

- Vonoprazan 10 mg

This multi-center observational survey will be conducted in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a history of gastric or duodenal ulcer

Exclusion Criteria:

* Participants with gastric or duodenal ulcer at initiation of vonoprazan therapy
* Participants with active upper gastrointestinal hemorrhage at initiation vonoprazan therapy
* Participants with a history of hypersensitivity to any ingredients in vonoprazan Tablets
* Participants receiving atazanavir sulfate or rilpivirine hydrochloride

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The survey population will consist of participants with a diagnosis of gastric or duodenal ulcers and during low-dose aspirin administration in the routine medical care.
Sampling Method: Probability Sample
Enrollment: 1119 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Takeda Selected Site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the survey at 121 investigative sites in Japan, from 01 September 2016 to 28 February 2019.
Pre-assignment Details: Participants with a historical diagnosis of gastric or duodenal ulcers were enrolled. Participants received vonoprazan as part of a routine medical care.
Period: Overall Study
Arm/Group | Vonoprazan 10 mg
Started | 1119
Completed | 1059
Not Completed | 60
Not completed — Case Report Forms Uncollected | 14
Not completed — Protocol Deviation | 46

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Arm/Group | Vonoprazan 10 mg
Number analyzed (Participants) | 1059
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.2 (10.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 309
  Male | 750
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants] — All participants were enrolled in Japan
  Participants
    Japan | 1059
Medical History [Count of Participants; unit: Participants] — Number of participants with or without medical history of Gastric Ulcer or Duodenal Ulcer was reported. Population: Participants could be counted in more than 1 category (including duplicates).
  Participants
    Gastric Ulcer | 946
    Duodenal Ulcer | 121
Purpose of Low-Dose Aspirin Use [Count of Participants; unit: Participants] — Population: Participants could be counted in more than 1 category (including duplicates).
  Participants
    Angina Pectoris | 464
    Myocardial Infarction | 278
    Transient Ischaemic Attack (TIA) Population | 27
    Cerebral Infarction | 294
    Others | 140
Implantation of Coronary Stent [Count of Participants; unit: Participants]
  Implanted | 484
  Not Implanted | 575
Healthcare Category [Count of Participants; unit: Participants] — Participants were categorized as outpatient and inpatient.
  Participants
    Outpatient | 695
    Inpatient | 364
Predisposition to Hypersensitivity [Count of Participants; unit: Participants] — Number of participants who had or did not have a liability or tendency to suffer from hypersensitivity was reported.
  Participants
    Had Predisposition to Hypersensitivity | 67
    Had No Predisposition to Hypersensitivity | 918
    Unknown | 74
Medical Complications [Count of Participants; unit: Participants] — Complications defined as a disease or a health condition for each participant at the start of study. Complications were classified as congenital anomalies, endocrine disorders, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, gastrointestinal (GI) disorders, renal disease and other complications. Other complications included all complications except for those mentioned above.
  Participants
    Had Medical Complications | 971
    Had No Medical Complications | 88
Height [Mean (Standard Deviation); unit: Centimeters (cm)] — Population: The number analyzed is the number of participants with data available for analysis.
  Centimeters (cm)
    number analyzed (Participants) | 927
    (all) | 160.52 (9.361)
Weight [Mean (Standard Deviation); unit: Kilograms (kg)] — Population: The number analyzed is the number of participants with data available for analysis.
  Kilograms (kg)
    number analyzed (Participants) | 949
    (all) | 61.92 (12.591)
BMI [Mean (Standard Deviation); unit: Kilogram (kg)/meter (m)^2] — Body Mass Index = weight (kg)/[height (m)^2] Population: The number analyzed is the number of participants with data available for analysis.
  Kilogram (kg)/meter (m)^2
    number analyzed (Participants) | 920
    (all) | 23.96 (3.710)
Helicobacter Pylori Infection [Count of Participants; unit: Participants] — Number of participants with or without medical history of H. pylori was reported.
  "Negative" indicates the absence of H. pylori infection, "Positive" indicates presence of the infection.
  Participants
    Helicobacter Pylori Positive | 16
    Helicobacter Pylori Negative | 107
    Unknown | 936
Smoking Classification [Count of Participants; unit: Participants]
  Never Smoked | 324
  Current Smoker | 136
  Ex-Smoker | 394
  Unknown | 205
Drinking Habits [Count of Participants; unit: Participants]
  Current Drinker | 226
  Never Drank or Ex Drinker | 537
  Unknown | 296
Presence of Stress as a Risk Factor of Gastric or Duodenal Ulcer [Count of Participants; unit: Participants]
  Present | 117
  Absent | 381
  Unknown | 561
Prior Treatment with Acid Suppressants to Prevent Recurrent Gastric or Duodenal Ulcer [Count of Participants; unit: Participants]
  Had Prior Treatment with Acid Suppressants | 507
  Had No Prior Treatment with Acid Suppressants | 529
  Unknown | 23

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Had One or More Adverse Drug Reactions
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. Adverse drug reaction refers to AE related to administered drug.
Time Frame: Up to 12 months
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Number; unit: Percentage of Participants
Arm/Group | Vonoprazan 10 mg
Number analyzed (Participants) | 1059
Percentage of Participants | 1.79

2. Secondary Outcome: Percentage of Participants With Gastric Ulcers After the Start of Administration of Vonoprazan Tablets
Description: Reported data were percentage of participants who experienced an onset of gastric ulcers after the start of administration of vonoprazan tablets.
Time Frame: Up to 12 months
Population: Efficacy assessment population, The efficacy assessment population was defined as participants who completed the survey and had efficacy data at baseline and post-baseline time points available.
Measure: Number; unit: Percentage of Participants
Arm/Group | Vonoprazan 10 mg
Number analyzed (Participants) | 1038
Percentage of Participants | 0.67

3. Secondary Outcome: Percentage of Participants With Duodenal Ulcers After the Start of Administration of Vonoprazan Tablets
Description: Reported data were percentage of participants who experienced an onset of duodenal ulcers after the start of administration of vonoprazan tablets.
Time Frame: Up to 12 months
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Vonoprazan 10 mg
Number analyzed (Participants) | 1038
Percentage of Participants | 0.19

4. Secondary Outcome: Percentage of Participants With Hemorrhagic Lesions on Stomach After the Start of Administration of Vonoprazan Tablets
Description: Reported data were percentage of participants who had hemorrhagic lesions on stomach after the start of administration of vonoprazan tablets.
Time Frame: Up to 12 months
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Vonoprazan 10 mg
Number analyzed (Participants) | 1038
Percentage of Participants | 0.19

5. Secondary Outcome: Percentage of Participants With Hemorrhagic Lesions on Duodenum After the Start of Administration of Vonoprazan Tablets
Description: Reported data were percentage of participants who had hemorrhagic lesions on duodenum after the start of administration of vonoprazan tablets.
Time Frame: Up to 12 months
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Vonoprazan 10 mg
Number analyzed (Participants) | 1038
Percentage of Participants | 0.00

ADVERSE EVENTS:
Time Frame: Up to 12 months
Description: At each visit the investigator had to document any occurrence of AEs and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to the survey treatment.
Arm/Group | Vonoprazan 10 mg
All-Cause Mortality (participants affected / at risk) | 9/1059
Serious Adverse Events (participants affected / at risk) | 50/1059
Other Adverse Events (participants affected / at risk) | 4/1059
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vonoprazan 10 mg (N=1059)
Endocarditis (Infections and infestations) | 1
Gangrene (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Sepsis (Infections and infestations) | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Carotid artery stenosis (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 1
Motor neurone disease (Nervous system disorders) | 1
Myelopathy (Nervous system disorders) | 1
Cataract nuclear (Eye disorders) | 1
Angina pectoris (Cardiac disorders) | 7
Angina unstable (Cardiac disorders) | 2
Atrioventricular block complete (Cardiac disorders) | 1
Heart failures (Cardiac disorders) | 3
Cardiac failure congestive (Cardiac disorders) | 2
Myocardial infarction (Cardiac disorders) | 1
Sinus node dysfunction (Cardiac disorders) | 1
Aortic aneurysm (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Cholangitis (Hepatobiliary disorders) | 2
Cholangitis acute (Hepatobiliary disorders) | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Vascular complication associated with device (General disorders) | 1
Vascular stent stenosis (General disorders) | 1
Angiocardiogram (Investigations) | 1
Shunt occlusion (Injury, poisoning and procedural complications) | 1
Shunt stenosis (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 0.3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vonoprazan 10 mg (N=1059)
Drug eruption (Skin and subcutaneous tissue disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2017-06-02): https://cdn.clinicaltrials.gov/large-docs/94/NCT03214094/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-07): https://cdn.clinicaltrials.gov/large-docs/94/NCT03214094/SAP_001.pdf